CLINICAL TRIAL: NCT07359469
Title: Evaluation of Intraoperative Intravenous Lidocaine, Ketamine, and Magnesium on Postoperative Pain and Opioid Use After Pulmonary Resection: A Prospective Observational Cohort Study
Brief Title: Intravenous Lidocaine, Ketamine, and Magnesium in Thoracic Surgery
Acronym: LKM-Thorax
Status: Completed | Type: Observational
Sponsor: Universidad Pública de Navarra (Other)
Responsible Party: Sponsor
Other Study IDs: FR-CP01; EDONA-UPNA-2025 (Other: Universidad Pública de Navarra (UPNA))
Record Dates: First submitted 2025-12-09; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Postoperative Pain; Thoracic Surgery; Multimodal Analgesia; Opioid Consumption, Postoperative
Keywords: Multimodal analgesia; Lidocaine; Ketamine; Magnesium sulphate; Opioid consumption; VAS pain score; thoracotomy; VATS surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lidocaine-Ketamine-Magnesium Group (LKM): Adult patients undergoing elective pulmonary resection who received intraoperative multimodal analgesia including continuous infusions of lidocaine, ketamine, and magnesium according to institutional protocol.
- Standard Analgesia Control Group: Adult patients undergoing elective pulmonary resection who received standard intraoperative analgesia without lidocaine, ketamine, or magnesium infusion.

SUMMARY:
Thoracic surgery often produces severe postoperative pain due to nerve injury and inflammation. Effective pain control is essential to reduce complications and opioid use. This prospective observational cohort study evaluated adult patients undergoing pulmonary resection by thoracotomy or video-assisted thoracoscopic surgery (VATS). The study examined whether intraoperative administration of intravenous lidocaine, ketamine, and magnesium, used as part of multimodal analgesia, was associated with reduced postoperative morphine consumption and lower early postoperative pain scores. Outcomes included 24-hour morphine use, pain intensity at 3 and 24 hours, complications, and chronic pain at 3 months. No study-directed interventions were performed; anesthetic management followed routine clinical practice.

DETAILED DESCRIPTION:
This prospective observational cohort study included 118 adult patients undergoing elective pulmonary resection between 2018 and 2022. The objective was to evaluate the association between intraoperative intravenous lidocaine, ketamine, and magnesium (LKM) and postoperative analgesic outcomes. Seventy-one patients received intraoperative LKM as part of a standardized multimodal analgesic protocol, consisting of lidocaine (1.5 mg/kg bolus followed by 1.5 mg/kg/h infusion), ketamine (0.3 mg/kg bolus), and magnesium sulfate (1.5 g bolus). Forty-seven patients received standard anesthesia without LKM administration. No study-specific interventions were assigned; exposure was based on routine anesthetic practice.

The primary outcome was total intravenous morphine consumption during the first 24 postoperative hours. Secondary outcomes included pain scores (VAS) at 3 and 24 hours, incidence of chronic postoperative pain at 3 months, pulmonary and cardiovascular complications, renal injury, thromboembolic events, hospital length of stay, and mortality. Safety monitoring included hypotension, bradycardia, arrhythmias, hallucinations, and delayed emergence from anesthesia.

This study aimed to identify perioperative factors influencing postoperative pain and opioid use after thoracic surgery, while evaluating the potential benefit of LKM within a multimodal analgesia strategy. All patients provided informed consent, and the study was approved by the local ethics committee. Data collection and clinical management followed standard institutional protocols.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Scheduled for elective pulmonary resection (thoracotomy or VATS).
* Able to provide informed consent.
* ASA physical status I-IV.

Exclusion Criteria:

* Emergency surgery.
* Known allergy or contraindication to lidocaine, ketamine, or magnesium.
* Severe hepatic insufficiency.
* Severe renal dysfunction (eGFR < 30 mL/min/1.73 m²).
* Pre-existing significant arrhythmias (e.g., uncontrolled atrial fibrillation, ventricular arrhythmias).
* Pregnancy.
* Cognitive impairment preventing valid informed consent.
* Patients receiving chronic intravenous analgesics or regional anesthesia techniques preoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective pulmonary resection (thoracotomy or video-assisted thoracoscopic surgery) at University Hospital Dr. Josep Trueta. The study population includes individuals receiving standard perioperative analgesic management and monitored in the postoperative care unit. Patients represent a typical thoracic surgery clinical population treated in routine practice.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Total intravenous morphine consumption within the first 24 hours postoperatively. | First 24 postoperative hours
  Total amount of intravenous morphine administered during the first 24 postoperative hours. Values will be recorded in milligrams (mg). Higher values indicate greater opioid consumption.

SECONDARY OUTCOMES:
Pain intensity at 3 and 24 hours postoperatively, assessed using a 10-point Visual Analogue Scale (VAS), chronic pain ( 3 months) | 3 hours, 24 hours, and 3 months after surgery
  Pain intensity assessed using a 10-point Visual Analogue Scale (VAS), where 0 represents no pain and 10 represents the worst imaginable pain. Measurements will be recorded at 3 hours, 24 hours, and 3 months after surgery. Higher scores indicate greater pain intensity. Pain persisting at 3 months will be classified as chronic post-surgical pain.

OTHER OUTCOMES:
Safety Outcomes | Perioperative period (day of surgery through postoperative day 7) and at 3 months
  Incidence of perioperative and postoperative adverse events, including hypotension, bradycardia, atrial fibrillation, deep vein thrombosis (DVT), pulmonary embolism (PE), prolonged hospital stay, in-hospital mortality, and survival status at 3 months. All events will be recorded as present or absent (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Murie Fernandez, MD, PhD, Principal Investigator — Universidad Pública de Navarra ( UPNA)
Locations (1):
- University Hospital Dr. Josep Trueta, Girona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study is observational and involves retrospective data collected as part of routine clinical care. Data cannot be shared publicly due to privacy and confidentiality restrictions.